CLINICAL TRIAL: NCT04590092
Title: Pessary Use for Stress Urinary Incontinence in Pregnancy: a Pilot Randomized Controlled Trial
Brief Title: Pessary Use for Stress Urinary Incontinence in Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Catherine Smith, Clinical Administrator, Advanced Training in Female Pelvic Medicine & Reconstructive Surgery (FPMRS) program, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H20-02900
Record Dates: First submitted 2020-09-29; First posted 2020-10-19 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Stress Urinary Incontinence; Pregnancy Related
Keywords: Stress urinary incontinence; Pregnancy; Pessary; Pelvic floor
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Study Participants who do not receive a pessary. This group will be given an information pamphlet on pelvic floor (Kegel) exercises in pregnancy and will continue to have standard antenatal care with their maternity provider.
- Pessary (Experimental): Study Participants who are fitted with a pessary for urinary incontinence. This group will be given an information pamphlet on pelvic floor (Kegel) exercises in pregnancy and pessary use in pregnancy. They will continue to have standard antenatal care with their maternity provider.
  Interventions: Device: Cooper Surgical Ring Pessary with Incontinence Knob

INTERVENTIONS:
Device: Cooper Surgical Ring Pessary with Incontinence Knob — A pessary is a silicone ring with a knob that in inserted into the vagina to treat urinary incontinence by providing urethral support.
  Arms: Pessary

SUMMARY:
When women are pregnant they are more likely to leak urine which can severely affect their quality of life. This problem could be fixed by using a pessary. A pessary is a silicone ring that goes into the vagina which can stop or improve urinary leakage. These devices have been safely used for hundreds of years. However, pessaries has not been studied for urinary leakage in pregnancy. The investigators would like to compare severity of urinary leakage using a number of questionnaires during the last 3 months of pregnancy for women using a pessary versus women without a pessary.

DETAILED DESCRIPTION:
Specific Aims To determine if an incontinence pessary will improve condition-specific quality of life for women with stress urinary incontinence (SUI) in the third trimester of pregnancy and collect pilot data to inform sample size and feasibility for a larger randomized controlled trial.

Background/Significance The prevalence of antenatal urinary incontinence (UI) in nulliparous women is 30-40%; the prevalence increases with multiparity and prior vaginal delivery. Stress urinary incontinence (SUI) and mixed urinary incontinence (MUI) are reported by 37% and 58% of gravidas respectively. Fifty percent of all new UI in pregnancy is SUI. As pregnancy progresses the prevalence of SUI increases from 8.3% to 36.9% in the third trimester. The frequency, volume and severity of the UI worsens with increasing gestational age, resulting in increasingly profound effects on women's daily life. These concerns are often underreported and under recognized by clinicians. SUI in pregnancy is currently managed with pelvic floor exercises, associated with incomplete symptom relief, suboptimal patient adherence and limited evidence.

Incontinence pessaries can be a ring or a dish with an incontinence knob. These pessaries decrease UI by providing compression and support to the urethra. Up to 63% of non-pregnant women fitted with an incontinence pessary are satisfied with the treatment at 3 months; after one year of use 50-59% of women remain satisfied and one third have "no bothersome SUI symptoms". Pessaries are a low risk and effective option to manage UI. The use of incontinence pessaries is supported for the treatment of SUI in non-pregnant women by the Society of Obstetrics and Gynaecology of Canada.

Pessaries are safe in pregnancy and have been reported for the management of cervical insufficiency, pelvic organ prolapse, and incarcerated uterus. While some believe pregnant women are ideal candidates for incontinence pessaries, supporting evidence is required. There are currently no obstetrical guidelines supporting pessary use for incontinence in pregnancy despite pessaries being a low risk treatment option; clinicians are currently limited to offering pelvic floor exercises for antepartum urinary incontinence. Pessaries are a safe and effective management option for UI in pregnancy and they can be managed independently by the patient.

Stress urinary incontinence represents a common concern in pregnancy and lacks evidence-based treatment options. In this pilot trial, the investigators propose to quantify the effect of incontinence pessaries on condition-specific quality of life and SUI symptoms in pregnant women, and to determine rate of successful pessary fitting, treatment acceptability, sexual function, patterns of adherence, discontinuation rate, adverse events and global impression of improvement. Our trial will provide important evidence for a much-needed larger clinical trial aiming to investigate incontinence pessaries as a treatment option for SUI in pregnancy.

Methodology

Design: Pilot randomized controlled trial

Sample Size: The effect size of a pessary for the treatment of SUI in pregnancy is unknown. A convenience sample of 60 women will be recruited, with 30 women randomized to the intervention arm (incontinence pessary) and 30 to the control arm (usual care).

Primary objective of pilot trial: To evaluate the effect size of an antepartum incontinence pessary on the condition-specific quality of life of women with SUI in pregnancy, in order to inform sample size calculations for a larger randomized controlled trial.

Secondary objectives of pilot trial: To evaluate feasibility and methodological barriers for a future randomized controlled trial.

Experimental Design:

The investigators propose a prospective randomized controlled pilot trial of women with bothersome SUI in the third trimester of a healthy singleton pregnancy. A convenience sample of 30 women per arm will be recruited from obstetrical clinics. Women between 26- 28weeks gestational age who answer yes to the screening question "Do you have bothersome urinary leakage when you cough, sneeze or walk during this pregnancy?" will be invited to participate in our proposed study by their primary maternity provider. The study coordinator will screen potential participants by phone to ensure they meet out inclusion and exclusion criteria and have a minimal Pelvic Floor Distress Inventory (PFDI-20) score of 25 for the UDI-6 section, to ensure bother from SUI. Informed consent will be obtained. Following recruitment, a baseline assessment (PFDI, Pelvic Floor Inventory Questionnaire (PFIQ), Female Sexual Function Inventory (FSFI) and a bladder diary) and collection of demographic data will be completed. These questionnaires will be emailed to participants. Participants will then be randomized to the control or treatment group. The control group will continue with standard obstetrical care while an incontinence pessary will be fitted for women in the treatment group by an experienced nurse incontinence advisor at our pessary clinic.

Following randomization all participants will be screened every two weeks from 28 weeks gestational age with the interim questionnaire. They will receive a biweekly phone call from either the nurse continence advisor or the urogynecology fellow. For the treatment arm this call will include their obstetric health, pessary tolerance and any adverse events. Women in the control group will be asked the interim obstetrical questions only. This will continue until delivery, pessary discontinuation, or 36 weeks gestational age at which point the patient will be discharged from the study. An exit interview will be completed and will consist of a final review of the biweekly questions, the questionnaires (PFDI, PFIQ, FSFI and a bladder diary), and the acceptability questionnaire for those participants using a pessary. Participants using a pessary will be asked to remove it at the end of the study. The investigators will also collect data on study feasibility including recruitment rate, methodological barriers, and follow up.

Intervention:

After deemed appropriate for recruitment, participants will be randomized to the control or intervention arm. Both groups will continue to receive routine antenatal care and will receive a handout on pelvic floor exercises in pregnancy. Women in the intervention arm will be fitted with an incontinence ring pessary by an incontinence nurse experienced in pessary fitting. They will be taught pessary maintenance and encouraged to remove and insert the pessary independently. Participants will receive a handout on pessary use, risks and obstetrical indications to remove the pessary.

Data Analysis:

Descriptive statistics on demographic characteristics will be reported. Condition-specific quality of life and distress scores will be compared between control and intervention arms using regression analysis adjusted for baseline score. Depending on the distribution of the data, linear, generalized linear or quantile regression will be used. The main analysis will be an intention-to-treat analysis which will include all women followed to the end of study, with sensitivity analysis being a per protocol analysis which excluded women who discontinued pessary prematurely. Effect size and variance will be calculated and used for future sample size calculations. Pessary fitting success rate, discontinuation rates, and adverse events will be continuously monitored. The investigators aim to recruit 2-3 women per week with a drop-out rate under 20%.

ELIGIBILITY:
Inclusion Criteria:

* English speaking women over 19 years old
* Nulliparous and multiparous women over 26 weeks gestational age with a healthy singleton pregnancy
* Bothersome symptoms of stress urinary incontinence or stress-predominant mixed urinary incontinence with a minimal PDFI score of 25 on the UDI-6 section.

Exclusion Criteria:

* Stage 3 or greater pelvic organ prolapse
* Contraindication to pessary use (known pelvic infection, vaginal or cervical lesions)
* Previous surgery for urinary incontinence
* History of preterm delivery and current threatened preterm labour
* Premature preterm rupture of membranes
* Short cervix
* Hospitalization in the current pregnancy
* Antepartum hemorrhage
* Fetal anomaly
* Prior trial of pessary or current pessary use
* Vulvodynia

Ages: 19 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
PFDI-20 score difference and variance | At exit interview (36 weeks gestational age)
  Pelvic Floor Disability Inventory (PFDI-20) score differences and variance between; intervention and control arms at 36 weeks gestational age; range 0-100; higher scores are a worse outcome.

SECONDARY OUTCOMES:
Pelvic Floor Impact Questionnaire (PFIQ-7) score | At exit interview (36 weeks gestational age)
  Differences between intervention and control arms; Rang 0-300, high scores are worse
Bladder Diary | At exit interview (36 weeks gestational age)
  Differences between intervention and control arms
Female Sexual Function Index (FSFI) score | At exit interview (36 weeks gestational age)
  Differences between intervention and control arms; Range 2-36; low scores have a worse outcome.
Pessary Usability | At exit interview (36 weeks gestational age)
  Patient acceptability and global impression questionnaire. Intervention arm only; Scale of 0-5; higher score means pessary is more acceptable.
Vaginal discharge | Biweekly from 28 weeks gestational age to 36 weeks gestational age
  Recorded as vaginal discharge present or absent
Pessary fitting and success | up to 24 months
  Number women with a successful fitting/total number of attempted fittings
evaluate study retention rates | up to 24 months
  number of women who leave the study before the formal discharge criteria are met
Abdominal Pain | Biweekly from 28 weeks gestational age to 36 weeks gestational age
  Recorded as abdominal pain present or absent
Pelvic pain | Biweekly from 28 weeks gestational age to 36 weeks gestational age
  Recorded as pelvic pain present or absent
Pessary expulsion | Biweekly from 28 weeks gestational age to 36 weeks gestational age
  Recorded as pessary has or has not fallen out of the vagina.
Incomplete emptying | Biweekly from 28 weeks gestational age to 36 weeks gestational age
  Recorded as incomplete emptying present or absent
Difficult removing pessary | Biweekly from 28 weeks gestational age to 36 weeks gestational age
  Recorded as the pessary is or is not difficult to remove.
Difficult inserting the pessary | Biweekly from 28 weeks gestational age to 36 weeks gestational age
  Recorded as the pessary is or is not difficult to insert.
Number of daily hours of pessary use | Biweekly from 28 weeks gestational age to 36 weeks gestational age
  Recorded as number of hours of pessary use on a daily bases.
Difficulty with sexual activity | Biweekly from 28 weeks gestational age to 36 weeks gestational age
  Recorded as yes or no difficulty with sexual activity
Vaginal Bleeding | Biweekly from 28 weeks gestational age to 36 weeks gestational age
  Recorded as absent or present.
Delivery | Biweekly from 28 weeks gestational age to 36 weeks gestational age
  Recorded as absent or present.
Hospital Admission | Biweekly from 28 weeks gestational age to 36 weeks gestational age
  Recorded as absent or present.
Group B strep Positive | Biweekly from 28 weeks gestational age to 36 weeks gestational age
  Recorded as absent or present.
Rupture of membranes | Biweekly from 28 weeks gestational age to 36 weeks gestational age
  Recorded as absent or present.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Smith, MD, Principal Investigator — University of British Columbia
Locations (1):
- Providence Health Care - St Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daly D, Clarke M, Begley C. Urinary incontinence in nulliparous women before and during pregnancy: prevalence, incidence, type, and risk factors. Int Urogynecol J. 2018 Mar;29(3):353-362. doi: 10.1007/s00192-018-3554-1. Epub 2018 Jan 23. PMID 29362836
- [Background] Balik G, Guven ES, Tekin YB, Senturk S, Kagitci M, Ustuner I, Mete Ural U, Sahin FK. Lower Urinary Tract Symptoms and Urinary Incontinence During Pregnancy. Low Urin Tract Symptoms. 2016 May;8(2):120-4. doi: 10.1111/luts.12082. Epub 2014 Dec 11. PMID 27111624
- [Background] Gyhagen M, Akervall S, Molin M, Milsom I. The effect of childbirth on urinary incontinence: a matched cohort study in women aged 40-64 years. Am J Obstet Gynecol. 2019 Oct;221(4):322.e1-322.e17. doi: 10.1016/j.ajog.2019.05.022. Epub 2019 May 21. PMID 31121136
- [Background] Brown SJ, Donath S, MacArthur C, McDonald EA, Krastev AH. Urinary incontinence in nulliparous women before and during pregnancy: prevalence, incidence, and associated risk factors. Int Urogynecol J. 2010 Feb;21(2):193-202. doi: 10.1007/s00192-009-1011-x. Epub 2009 Oct 16. PMID 19834637
- [Background] Solans-Domenech M, Sanchez E, Espuna-Pons M; Pelvic Floor Research Group (Grup de Recerca del Sol Pelvia; GRESP). Urinary and anal incontinence during pregnancy and postpartum: incidence, severity, and risk factors. Obstet Gynecol. 2010 Mar;115(3):618-628. doi: 10.1097/AOG.0b013e3181d04dff. PMID 20177295
- [Background] Robert M, Schulz JA, Harvey MA; UROGYNAECOLOGY COMMITTEE. RETIRED: Technical update on pessary use. J Obstet Gynaecol Can. 2013 Jul;35(7):664-674. doi: 10.1016/S1701-2163(15)30888-4. PMID 23876646
- [Background] Richter HE, Burgio KL, Brubaker L, Nygaard IE, Ye W, Weidner A, Bradley CS, Handa VL, Borello-France D, Goode PS, Zyczynski H, Lukacz ES, Schaffer J, Barber M, Meikle S, Spino C; Pelvic Floor Disorders Network. Continence pessary compared with behavioral therapy or combined therapy for stress incontinence: a randomized controlled trial. Obstet Gynecol. 2010 Mar;115(3):609-617. doi: 10.1097/AOG.0b013e3181d055d4. PMID 20177294
- [Background] Farrell SA, Singh B, Aldakhil L. Continence pessaries in the management of urinary incontinence in women. J Obstet Gynaecol Can. 2004 Feb;26(2):113-7. doi: 10.1016/s1701-2163(16)30486-8. PMID 14965476
- [Background] Geoffrion R, Zhang T, Lee T, Cundiff GW. Clinical characteristics associated with unsuccessful pessary fitting outcomes. Female Pelvic Med Reconstr Surg. 2013 Nov-Dec;19(6):339-45. doi: 10.1097/SPV.0b013e3182a26174. PMID 24165447
- [Background] Vasconcelos CTM, Silva Gomes ML, Ribeiro GL, Oria MOB, Geoffrion R, Vasconcelos Neto JA. Women and healthcare providers' knowledge, attitudes and practice related to pessaries for pelvic organ prolapse: A Systematic review. Eur J Obstet Gynecol Reprod Biol. 2020 Apr;247:132-142. doi: 10.1016/j.ejogrb.2020.02.016. Epub 2020 Feb 14. PMID 32113060
- [Background] Saccone G, Ciardulli A, Xodo S, Dugoff L, Ludmir J, Pagani G, Visentin S, Gizzo S, Volpe N, Maruotti GM, Rizzo G, Martinelli P, Berghella V. Cervical Pessary for Preventing Preterm Birth in Singleton Pregnancies With Short Cervical Length: A Systematic Review and Meta-analysis. J Ultrasound Med. 2017 Aug;36(8):1535-1543. doi: 10.7863/ultra.16.08054. Epub 2017 Apr 11. PMID 28398701
- [Background] Jarde A, Lutsiv O, Beyene J, McDonald SD. Vaginal progesterone, oral progesterone, 17-OHPC, cerclage, and pessary for preventing preterm birth in at-risk singleton pregnancies: an updated systematic review and network meta-analysis. BJOG. 2019 Apr;126(5):556-567. doi: 10.1111/1471-0528.15566. Epub 2018 Dec 29. PMID 30480871
- [Background] Zeng C, Yang F, Wu C, Zhu J, Guan X, Liu J. Uterine Prolapse in Pregnancy: Two Cases Report and Literature Review. Case Rep Obstet Gynecol. 2018 Oct 22;2018:1805153. doi: 10.1155/2018/1805153. eCollection 2018. PMID 30425870
- [Background] De Vita D, Giordano S. Two successful natural pregnancies in a patient with severe uterine prolapse: A case report. J Med Case Rep. 2011 Sep 14;5:459. doi: 10.1186/1752-1947-5-459. PMID 21917162
- [Background] Rusavy Z, Bombieri L, Freeman RM. Procidentia in pregnancy: a systematic review and recommendations for practice. Int Urogynecol J. 2015 Aug;26(8):1103-9. doi: 10.1007/s00192-014-2595-3. Epub 2015 Jan 20. PMID 25600351
- [Background] Yohannes P, Schaefer J. Urinary retention during the second trimester of pregnancy: a rare cause. Urology. 2002 Jun;59(6):946. doi: 10.1016/s0090-4295(02)01551-0. PMID 12031388
- [Background] Viera AJ, Larkins-Pettigrew M. Practical use of the pessary. Am Fam Physician. 2000 May 1;61(9):2719-26, 2729. PMID 10821152
- [Background] Al-Shaikh G, Syed S, Osman S, Bogis A, Al-Badr A. Pessary use in stress urinary incontinence: a review of advantages, complications, patient satisfaction, and quality of life. Int J Womens Health. 2018 Apr 17;10:195-201. doi: 10.2147/IJWH.S152616. eCollection 2018. PMID 29713205